CLINICAL TRIAL: NCT01181817
Title: Evaluation of the Brain Activity During Spinal Cord Stimulation (SCS) in Failed Back Surgery Syndrome Using Functional Magnetic Resonance Imaging (fMRI) and Magnetic ResonanceSpectroscopy (MRS)
Brief Title: Evaluation of the Brain Activity During Spinal Cord Stimulation in Failed Back Surgery Syndrome Using Functional MRI and MRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Maarten Moens (Unknown)
Responsible Party: Maarten Moens, MD, Neurosurgery
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: vubmtmoensSCS
Record Dates: First submitted 2010-08-10; First posted 2010-08-13 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2008-09

CONDITIONS: Failed Back Surgery Syndrome
Keywords: FBSS; at least one prior spinal surgery
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SCS (Other): patients with Failed back Surgery syndrome treated with SCS
  Interventions: Other: fMRI and MRS

INTERVENTIONS:
Other: fMRI and MRS — fMRI and MRS

SUMMARY:
Functional Magnetic Resonance Imaging (fMRI)and MR Spectroscopy of the brain are perfect tools to investigate the changes in the brainstem and brain evoked by the orthodromically impulses of a SCS.

DETAILED DESCRIPTION:
In case a patient meets all inclusion and no exclusion criteria, he/she will be implanted with an epidural neurostimulation lead (electrode).

The day of implant will be recorded as day 0 (table 1) and will always be a Thursday.

Post lead implant, the patient will be hospitalized for a small week as per common practice in case of the intervention outside of the study.

During hospital stay, the investigator of the study, or a representative of the product manufacturer, Medtronic®, will search for the optimal stimulation parameters to evoke correct paraesthesia coverage and pain relief. If appropriate parameters have been found, these will be saved in the external neurostimulator.

After maximum one hour, the neurostimulator will be turned off again.

On day 12, a Tuesday, a MR spectrospoy will be performed. Each patient will undergo three sessions.

Each session will be divided into a MR spectroscopy session and fMRI session without stimulation and a session with stimulation. The MR spectroscopy session without stimulation will bring us the baseline in neurobiology of neuropathic pain; after measurement, the stimulator will be switch on and a MR spectroscopy will be performed during a longer period of time (10 min) in order to determine neurobiological changes in time during SCS.

The 3 MR spectroscopy sessions will be performed on different regions in the brain (both talami and rostral region of anterior cingulated cortex)

ELIGIBILITY:
Inclusion Criteria:

1. Age male/female patient ≥ 18 years
2. Patient diagnosed with Failed Back Surgery Syndrome with at least one prior spinal surgery
3. Patient with low back pain and/or pain in at least one leg
4. Pain intensity at baseline assessed by VAS > 5 (50%)
5. Patient willing to provide informed consent.

Exclusion Criteria:

1. Use of spinal cord stimulation in this patient in the past.
2. Presence of other clinically significant or disabling chronic pain condition
3. Expected inability of patients to receive or properly operate the spinal cord stimulation system
4. History of coagulation disorders, lupus erythematosus, diabetic neuropathy, rheumatoid arthritis or morbus Bechterew
5. Active malignancy
6. Current use of medication affecting coagulation which cannot be temporarily stopped
7. Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by investigator
8. Life expectancy of less than 1 year
9. Existing or planned pregnancy
10. Existing extreme fear for entering MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
functional and neurobiological cerebral changes due to SCS | 2 years
  To compare brain activity before and after spinal cord stimulation (with appropriate paraesthesia) using functional magnetic resonance imaging and neurobiological changes in the spectrum (gamma-aminobutyric acid (GABA) glutamate (Glu) glutamine (Gln) N-acetylaspartate (NAA) Choline-containing compounds (Cho) Creatine plus phophocreatine (total creatine: Cr) Myo-inositiol (Ins) Choline (Cho) Glucose (Glc) Lactate (Lac)) due to stimulation measured by MRS. The primary outcome is the difference in neurobiology between baseline and when the stimulator is on.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Brussels Capital, Belgium